CLINICAL TRIAL: NCT04397042
Title: Evaluation of Signal Peptide, Complement C1r/C1s, Uegf, and Bmp1 (CUB), and Epidermal Growth Factor-like Domain-containing Protein-1(SCUBE-1) Levels and Carotid Intima-Media Thickness in Unexplained Recurrent Pregnancy Loss
Brief Title: SCUBE-1 and Carotid Intima Media Thickness in Recurrent Pregnancy Loss
Status: Suspended | Type: Observational
Why Stopped: pandemic
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sabri Colak, Asst. Prof. Sabri Colak,Department of Obstetrics and Gynecology, Recep Tayyip Erdogan University School of Medicine, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Recurrent Pregnancy Loss
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Pregnancy Loss
Keywords: recurrent pregnancy loss; unexplained; SCUBE-1; Carotis Intima-Media Thickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- recurrent pregnancy loss: Group 1 included thirty women admitted to our clinic for termination of pregnancy due to absence of fetal cardiac activity or absence of fetal pole on ultrasonographic examination. Patients with a history of two or more unexplained first trimester miscarriages and no live births were included in the study

SUMMARY:
Clinical research will be carried out on two groups of patients. It will be performed on people with recurrent pregnancy loss and without a history of pregnancy loss. In two groups, blood samples will be assessed by elisa test, SCUBE-1 level and carotis intima media thickness will be evaluated by ultrasonographic measurement. It will be investigated whether there is a statistically significant difference between the two groups.A statistically significant difference in SCUBE-1 and carotid intima media thickness known as ischemia markers is expected in the group with recurrent pregnancy loss that could not be explained in the hypothesis of this planned study.

DETAILED DESCRIPTION:
A total of 80 women who will apply to our obstetric clinic for early pregnancy loss or routine first trimester prenatal care will be included in the study. Patients will be divided into two groups. In Group 1, 40 women who applied to our clinic will be included due to the absence of fetal cardiac activity or fetal pole in ultrasonographic examination. Patients with two or more unexplained first trimester abortions and no live births will be included in the study. Pregnancies in the first trimester will be excluded. Group 2 will include 40 consecutive healthy women with at least one uneventful natural pregnancy for prenatal care in the first trimester. Women with normal pregnancy outcomes and no previous pregnancy loss will be included in the study. Patients who previously had diabetes or vascular disease will be excluded. The result of healthy pregnancy will be defined as delivery after 37 weeks, where the newborn birth weight was above the 10th percentile for pregnancy and no hypertensive or diabetic disease of pregnancy.

The gestational age for patients in the control group was calculated from the last menstrual period and will be verified by ultrasound examinations performed during the recording by trained ultrasonographers. It will be performed in the recurrent pregnancy loss (RPL) group according to the last menstrual period and previous sonography records of existing pregnancies without an existing fetal pole or intrauterine death. All results of term pregnancies for group 2, will be checked by reviewing the main delivery suit database and individual patient records A research protocol will be carried out to exclude known RPL relationships, such as antiphospholipid syndrome (APS) and an approved genetic abnormality. Recurrent abortions will include testing blood for diabetes, thyroid problems, autoimmune antibodies, coagulation factors, and parental karyotypes, and previous hysterosalpingography for abnormal uterine cavity. All couples diagnosed with chromosomal, anatomical, endocrinological and autoimmunological etiology of recurrent pregnancy loss will be excluded from group 1. Women with a history of ischemic disease, diabetes, heart disease, hypertension, or any known medical condition will not be recorded in two groups. Multiple pregnancy, any major or minor fetal anomaly, or existing smokers will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

Patients with a history of two or more unexplained first trimester miscarriages Healthy women attending for antenatal care with at least one previous uneventful natural pregnancy.

Women with normal pregnancy outcome and no previous pregnancy loss.

Exclusion Criteria:

No occurrence of hypertensive or diabetic disease of pregnancy. Pregnancies beyond the first trimester will be excluded from the study Pre-existing diabetes Vascular disease Antiphospholipid syndrome (APS) Genetic abnormality(chromosomal anomaly) Anatomic disorder Endocrinologic disorder Autoimmunologic disorder Ischemic diseases Diabetes mellitus Heart disease Hypertension Medical condition Multiple pregnancy Fetal anomaly current smokers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted with the patients admitted to the obstetric and gynecologic clinic of Recep Tayyip Erdogan University Hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-11-22 (Estimated); Study Completion 2022-06-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the levels of scube1 in patients with recurrent pregnancy loss | baseline
  Serum samples will be taken from all study group members. The study will be conducted with the given samples after routine assessment. 5 mL of maternal blood will be collected from the vein into tube, to be centrifuged within 1 h at 1000 g for 15 min. The plasma will be separated and stored at -80'C for analysis. Serum levels of SCUBE-1 will be quantified by ELISA using commercially available matched antibodies.

SECONDARY OUTCOMES:
Measurement of carotis intima media thickness by ultrasonography in recurrent pregnancy patients | baseline
  A high-resolution 7.5 megahertz (MHz) linear array ultrasound transducer (Hitachi 6500) will be used to measure Carotid Intima-Media Thickness (CIMT). It will be measured from the far wall of the right carotid artery within 10 mm proximal to the bifurcation on two-dimensional ultrasound images. Three points will be measured on 1 scan, synchronized with the R-wave peaks on the ECG to avoid possible errors resulting from variable arterial compliance. Mean CIMT will be calculated from 6 measurements on 2 scans. Measurements will be repeated 2 days later in 10 control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: sabri colak, Asst.Prof., Study Chair — faculty of medicine recep tayyip erdogan university
Locations (1):
- Recep Tayyip Erdogan University Faculty of Medicine, Department ofDepartment of Obstetrics and Gynecology, Rize, Turkey (Türkiye)

REFERENCES:
- [Background] Stephenson MD. Frequency of factors associated with habitual abortion in 197 couples. Fertil Steril. 1996 Jul;66(1):24-9. PMID 8752606
- [Background] Greenwold N, Jauniaux E, Gulbis B, Hempstock J, Gervy C, Burton GJ. Relationship among maternal serum endocrinology, placental karyotype, and intervillous circulation in early pregnancy failure. Fertil Steril. 2003 Jun;79(6):1373-9. doi: 10.1016/s0015-0282(03)00364-9. PMID 12798885
- [Background] Tu CF, Yan YT, Wu SY, Djoko B, Tsai MT, Cheng CJ, Yang RB. Domain and functional analysis of a novel platelet-endothelial cell surface protein, SCUBE1. J Biol Chem. 2008 May 2;283(18):12478-88. doi: 10.1074/jbc.M705872200. Epub 2008 Feb 26. PMID 18303018
- [Background] Xavier GM, Economou A, Senna Guimaraes AL, Sharpe PT, Cobourne MT. Characterization of a mouse Scube3 reporter line. Genesis. 2010 Dec;48(12):684-92. doi: 10.1002/dvg.20678. Epub 2010 Nov 19. PMID 20957652
- [Background] Dai DF, Thajeb P, Tu CF, Chiang FT, Chen CH, Yang RB, Chen JJ. Plasma concentration of SCUBE1, a novel platelet protein, is elevated in patients with acute coronary syndrome and ischemic stroke. J Am Coll Cardiol. 2008 Jun 3;51(22):2173-80. doi: 10.1016/j.jacc.2008.01.060. PMID 18510966
- [Background] Mensah GA. Healthy endothelium: the scientific basis for cardiovascular health promotion and chronic disease prevention. Vascul Pharmacol. 2007 May;46(5):310-4. doi: 10.1016/j.vph.2006.10.013. Epub 2006 Nov 21. PMID 17229594
- [Background] Altin C, Yilmaz M, Ozsoy HM, Gezmis E, Balci S, Tekindal MA, Sade LE, Muderrisoglu H. Assessment of epicardial fat and carotid intima media thickness in gestational hypertension. J Obstet Gynaecol Res. 2018 Jun;44(6):1072-1079. doi: 10.1111/jog.13631. Epub 2018 Mar 30. PMID 29603491
- [Background] Carpenter M, Sinclair H, Kunadian V. Carotid Intima Media Thickness and Its Utility as a Predictor of Cardiovascular Disease: A Review of Evidence. Cardiol Rev. 2016 Mar-Apr;24(2):70-5. doi: 10.1097/CRD.0000000000000077. PMID 26825762
- [Background] Lamarca B. The role of immune activation in contributing to vascular dysfunction and the pathophysiology of hypertension during preeclampsia. Minerva Ginecol. 2010 Apr;62(2):105-20. PMID 20502423
- [Background] Prefumo F, Gaze DC, Papageorghiou AT, Collinson PO, Thilaganathan B. First trimester maternal serum ischaemia-modified albumin: a marker of hypoxia-ischaemia-driven early trophoblast development. Hum Reprod. 2007 Jul;22(7):2029-32. doi: 10.1093/humrep/dem095. Epub 2007 Apr 16. PMID 17437959